CLINICAL TRIAL: NCT05379231
Title: Evaluate the Benefit of a BiCROS Hearing Aid Fitting
Brief Title: Evaluation of BiCROS Fitting Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 461
Record Dates: First submitted 2022-04-08; First posted 2022-05-18 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2023-03

CONDITIONS: Unilateral Deafness
MeSH Terms: conditions — Hearing Loss, Unilateral

STUDY DESIGN:
Intervention Model Description: All participants were wearing the BiCROS fitting during home trial, and tested in-lab with all conditions, randomized and counterbalanced (BiCROS fitting, monaural fitting, unaided).
Masking Description: Participants were wearing the BiCROS fitting during home trial, where no masking was possible. For in-lab tests, the CROS device was deactivated for the monaural condition, allowing for some masking. The unaided condition could not be masked. Participants were not aware which beamformer configuration was active during in-lab tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- BiCROS fitting with beamformer (Experimental): Each participant will be fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear. A beamformer (directional microphone) will be enabled during this measurement. Although each ear receives a different device configuration depending on the condition, the participant is assigned as a whole, and assignment is not by ears.
  Interventions: Device: Hearing aid fitting
- BiCROS fitting omni (Experimental): Each participant will be fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear. The microphones will be omnidirectional. Although each ear receives a different device configuration depending on the condition, the participant is assigned as a whole, and assignment is not by ears.
  Interventions: Device: Hearing aid fitting
- Monaural hearing aid fitting with beamformer (Active Comparator): Each participant will be fitted with a hearing aid on the better hearing ear and no device on the unaidable ear. A beamformer (directional microphone) will be enabled during the measurement. Although each ear receives a different device configuration depending on the condition, the participant is assigned as a whole, and assignment is not by ears.
  Interventions: Device: Hearing aid fitting
- Monaural hearing aid fitting omni (Active Comparator): Each participant will be fitted with a hearing aid on the better hearing ear and no device on the unaidable ear. The microphone will be omnidirectional. Although each ear receives a different device configuration depending on the condition, the participant is assigned as a whole, and assignment is not by ears.
  Interventions: Device: Hearing aid fitting
- Unaided condition (No Intervention): No intervention, the participants are not fitted with a CROS device and/or hearing aid.

INTERVENTIONS:
Device: Hearing aid fitting — A participant will wear a hearing aid with and without a CROS device on the unaidable ear.
  Arms: BiCROS fitting omni; BiCROS fitting with beamformer; Monaural hearing aid fitting omni; Monaural hearing aid fitting with beamformer

SUMMARY:
22 candidates for BiCROS hearing aids will be recruited and fitted with a hearing aid and a CROS device. Following a real-world trial, each participant will be tested on a range of outcome measures including speech recognition in noise, ratings of listening effort, and ratings of preference.

DETAILED DESCRIPTION:
Unilateral Hearing Loss (UHL) can be defined as any degree of permanent hearing loss on one ear with normal hearing in the opposite ear. Unilateral hearing loss can be debilitating associated with audiological, psychosocial and educational challenges. Audiological challenges include the reduced ability to localize sounds, reduced awareness on the unaidable side and difficulties hearing in noise or at a distance.

One solution for unaidable UHL is Contralateral Routing of Signals (CROS) and Bilateral Contralateral routing of signals (BiCROS) using a so-called CROS transmitter together with a hearing aid.

The rationale for this clinical investigation is to collect clinical data with a rechargeable CROS transmitter to evaluate the benefits of a BiCROS fitting compared to the alternative treatment option, the monaural hearing aid fitting, and to no treatment in noisy listening situations.

Hearing tests, ear impressions and hearing aid fitting visits are mainly conducted at the National Centre for Audiology in London, Ontario. Those visits are available at the Sonova Innovation Centre Toronto in Mississauga, Ontario, upon request. Outcome measurements are only conducted at the National Centre for Audiology in London, Ontario.

ELIGIBILITY:
Inclusion Criteria:

* unaidable hearing loss in worse ear (>N6)
* aidable hearing loss (N3 to N5) on the other ear
* fluent English speaker

Exclusion Criteria:

- aidable hearing loss in both ears

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Scollie, Principal Investigator — Western University, Canada
Locations (2):
- Canada (2):
  - National Centre for Audiology, London, Ontario
  - Sonova Innovation Centre Toronto, Mississauga, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants had to be excluded from continuing in the study before assignment because they did not meet the inclusion criteria.
Groups:
- Complete Sample: All participants first underwent a Home Visit where they all received a BiCROS fitting in the automatic mode, and then underwent an in-lab visit where all participants were randomized and counter-balanced into receiving 5 interventions (BiCROS Fitting with beamformer, BiCROS Fitting Omni, Monaural Fitting with Beamformer, Monaural Fitting Omni, and Unaided) in a different order/sequence.
  BiCROS fitting with beamformer: fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear. A beamformer will be enabled during this measurement.
  BiCROS fitting omni: fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear. The microphones will be omnidirectional.
  Monaural hearing aid fitting with beamformer: fitted with a hearing aid on the better hearing ear and no device on the unaidable ear. A beamformer will be enabled during the measurement.
  Monaural hearing aid fitting omni: fitted with a hearing aid on the better hearing ear and no device on the unaidable ear. The microphone will be omnidirectional.
  Unaided condition: No intervention, the participants are not fitted with a CROS device and/or hearing aid.
Period: Home Visit
Arm/Group | Complete Sample
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: In-lab Visit
Arm/Group | Complete Sample
Started | 20
BiCROS Fitting With Beamformer | 20
BiCROS Fitting Omni | 20
Monaural Hearing Aid Fitting With Beamformer | 20
Monaural Hearing Aid Fitting Omni | 20
Unaided Condition | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Complete Sample: All participants will perform the same tests in all conditions. Although each ear receives a different device configuration depending on the condition, the participant is assigned as a whole, and assignment is not by ears.
  BiCROS fitting: Each participant will be fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear.
  Monaural hearing aid fitting: Each participant will be fitted with a hearing aid on the better hearing ear and no device on the unaidable ear.
  Unaided condition: No intervention, the participants are not fitted with a CROS device and/or hearing aid.
  Since the characteristics of each "arm" are unrelevant for the study outcome, there has been no separate analysis on each "arm".
Arm/Group | Complete Sample
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: years] | 74.6 [61 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 18
BiCROS fitting candidate [Count of Participants; unit: Participants] | 18

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility in Noise Measured With US Matrix Test (Noise From a Defined Loudspeaker)
Description: Measuring the Signal to Noise Ratio change in decibels (dB) for speech from the front loudspeaker and noise from the better ear's side with the US matrix Test. Results of the speech test will be the SRT (speech recognition threshold) in dB SNR (signal to noise ratio).
  The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A)).
  The noise will be presented on the better ear at an azimuth of 90° or 270° (depending on the site of the better ear), at a level of 65 dB (A).
Time Frame: At the appointment following the 4 weeks home trial each participant went on wearing the BiCROS fitting
Population: Although each ear receives a different device configuration depending on the condition (except for the unaided condition), the participant is assigned as a whole, and assignment is not by ears.
Measure: Mean (Standard Deviation); unit: dBSRT
Groups:
- BiCROS With Beamformer: Each participant will be fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear. A beamformer (directional microphone) will be enabled during this measurement.
- BiCROS Omni: Each participant will be fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear. The microphones will be omnidirectional.
- Monaural With Beamformer: Each participant will be fitted with a hearing aid on the better hearing ear and no device on the unaidable ear. A beamformer (directional microphone) will be enabled during the measurement.
- Monaural Omni: Each participant will be fitted with a hearing aid on the better hearing ear and no device on the unaidable ear. The microphone will be omnidirectional.
- Unaided: No hearing aid fitting.
Arm/Group | BiCROS With Beamformer | BiCROS Omni | Monaural With Beamformer | Monaural Omni | Unaided
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
dBSRT | -8.8 (3.4) | -3.7 (2.9) | -9.2 (2.7) | -2.8 (2.5) | -0.1 (6.8)

2. Secondary Outcome: Speech Intelligibility in Noise Measured With US Matrix Test (Diffuse Noise)
Description: Measuring the Signal to Noise Ratio change in decibels (dB) for speech from the front loudspeaker in surrounding noise with the US Matrix Test. Results of the speech test will be the SRT (speech recognition threshold) in dB SNR (signal to noise ratio).
  The target speaker will be presented from 0° azimuth and is adaptive (start level at 65dB (A).
  The noise will be presented from a circle of 8 surrounding speakers from 45° to 315° at a level of 65 dB (A) with the participant seated in the centre of the circle.
Time Frame: At the appointment following the 4 weeks home trial each participant went on wearing the BiCROS fitting
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dBSRT
Arm/Group | BiCROS With Beamformer | BiCROS Omni | Monaural With Beamformer | Monaural Omni | Unaided
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
dBSRT | -14.2 (3.3) | -8 (4.2) | -13.9 (3.6) | -9.3 (3) | -3.4 (9.4)

3. Secondary Outcome: Reports of Subjective Quality of Hearing as Assessed by the SSQ
Description: Measured after home trial with the Speech, Spatial and Qualities of Hearing Scale-Benefit (Gatehouse, 2004). The scale ranges from -5 to 5, where negative values indicate that the condition under test is worse than the comparator, 0 indicates no change, and positive values indicate a benefit of the condition under test compared to the comparator.
Time Frame: At the appointment following the 4 weeks home trial each participant went on wearing the BiCROS fitting
Population: Although each ear receives a different device configuration, the participant is assigned as a whole, and assignment is not by ears.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BiCROS: Each participant will be fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear and wear the devices in automat during the home trial.
Arm/Group | BiCROS
Number analyzed (Participants) | 18
score on a scale
  Speech | 2.48 (0.59)
  Spatial | 1.16 (0.47)
  Qualities | 2.55 (0.35)

4. Secondary Outcome: Reports of Subjective Quality of Hearing as Assessed by the Bern Benefit Questionnaires
Description: Measured after home trial with the Bern Benefit in Single-Sided Deafness Questionnaire (Komps et al, 2011). The scale ranges from -5 to 5, where negative values indicate that the condition under test is better wihtout the hearing aid, 0 indicates no change, and positive values indicate a benefit with the hearing aid.
Time Frame: At the appointment following the 4 weeks home trial each participant went on wearing the BiCROS fitting
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiCROS
Number analyzed (Participants) | 18
score on a scale | 2.83 (0.76)

5. Secondary Outcome: Sound Quality Ratings for Total Impression and Clarity Using Gabriellson et al (1990) Ratings Scales
Description: Ratings of speech in noise presented via loudspeakers using Gabriellson et al (1990) Ratings Scales. Scales include Clarity and Total Impression, and range from 1 to 10. The higher the rating, the better the Clarity and Total Impression.
Time Frame: At the appointment following the 4 weeks home trial each participant went on wearing the BiCROS fitting
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiCROS With Beamformer | BiCROS Omni | Monaural With Beamformer | Monaural Omni | Unaided
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
score on a scale
  Clarity | 6.8 (2.4) | 5.2 (2.8) | 6.5 (2.3) | 4.8 (2.8) | 3.7 (3)
  Total Impression | 6.1 (2.7) | 4.7 (2.8) | 6 (2.3) | 4.3 (2.5) | 3.7 (2.6)

6. Secondary Outcome: Subjective Preference of Hearing Aid Condition
Description: 3 alternative forced choice (A, B, no preference or ABX) paradigm with three repetitions for speech in noise presented via loudsepakers
Time Frame: At the appointment following the 4 weeks home trial each participant went on wearing the BiCROS fitting
Measure: Count of Participants; unit: Participants
Groups:
- BiCROS w/ Beamformer vs. Monaural w/ Beamformer: Microphones of both fitting conditions were set to directional. Count indicates which fitting configuration participants preferred.
- BiCROS Omni vs. Monaural Omni: Microphones of both fitting conditions were set to omnidirectional. Count indicates which fitting configuration participants preferred.
- BiCROS Omni vs. w/ Beamformer: Omnidirectional and directional BiCROS fittings are compared. Count indicates which fitting configuration participants preferred.
- Monaural Omni vs. w/ Beamformer: Omnidirectional and directional monaural fittings are compared. Count indicates which fitting configuration participants preferred.
Arm/Group | BiCROS w/ Beamformer vs. Monaural w/ Beamformer | BiCROS Omni vs. Monaural Omni | BiCROS Omni vs. w/ Beamformer | Monaural Omni vs. w/ Beamformer
Number analyzed (Participants) | 18 | 18 | 18 | 18
Participants
  No preference | 7 | 11 | 2 | 4
  Monaural | 6 | 3 | 0 | 0
  BiCROS | 5 | 4 | 0 | 0
  Directional | 0 | 0 | 16 | 14
  Omnidirectional | 0 | 0 | 0 | 0

7. Secondary Outcome: Listening Effort in Noise Using 7 Point Scale (Holmes et. al., 2018)
Description: Measuring listening effort for speech in multi-talker babble presented via loudspeaker. The scale ranges from 1 to 7, and a higher rating indicates less listening effort.
Time Frame: At the appointment following the 4 weeks home trial each participant went on wearing the BiCROS fitting
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BiCROS With Beamformer | BiCROS Omni | Monaural With Beamformer | Monaural Omni | Unaided
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
score on a scale | 3.75 (1.8) | 4.9 (1.9) | 3.9 (1.6) | 5 (1.5) | 5.7 (1.8)

ADVERSE EVENTS:
Time Frame: From the first appointment the participant was enrolled and assessed, until the last appointment that concluded the home trial and study participation. The whole duration was about 5-6 weeks per participant.
Description: Studies involving the trial of a hearing aid are usually classified as low risk studies with low probability for serious adverse events or all-cause mortality.
Groups:
- Complete Sample: All participants will perform the same tests in all conditions. The order of the conditions is randomized but will be performed in the same visit by each participant. Although each ear receives a different device configuration depending on the condition, the participant is assigned as a whole, and assignment is not by ears.
  BiCROS fitting: Each participant will be fitted with the experimental CROS device on the unaidable ear and with a compatible hearing aid on the other ear.
  Monaural hearing aid fitting: Each participant will be fitted with a hearing aid on the better hearing ear and no device on the unaidable ear.
  Unaided condition: No intervention, the participants are not fitted with a CROS device and/or hearing aid.
  Since all participants wore the same condition for the home trial and performed testing with all conditions in the appointment afterwards, Adverse Events are not reported by different arms.
Arm/Group | Complete Sample
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complete Sample (N=22)
Ear infection (Ear and labyrinth disorders) | 1 (1) — Patient has had ear infections in the past (prior to study commencement). Developed a bilateral ear infection in the past week and had visited their physician for it.
Early withdrawal (unrelated) (Surgical and medical procedures) | 1 (1) — Participant decided to withdraw from study for health reasons unrelated to the investigational device or study procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT05379231/Prot_SAP_000.pdf